CLINICAL TRIAL: NCT03631212
Title: An Avatar-led Acceptance and Commitment Therapy Intervention Promotes Smoking Cessation in Young Adults
Brief Title: Avatar-led Acceptance and Commitment Therapy Smoking Cessation
Acronym: Flexiquit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Maria Karekla, Assistant Professor, University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ΕΕΒΚ/ΕΠ/2013/05
Record Dates: First submitted 2018-08-07; First posted 2018-08-15 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Smoking Cessation
Keywords: virtual humans; smoking cessation; youth; digital intervention; Acceptance and Commitment Therapy
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Comparison between flexiquit and a wait-list control group
Masking Description: No masking was carried out
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control (No Intervention): Wait-list control group
- Flexiquit (Experimental): Digital ACT-based intervention for smoking cessation
  Interventions: Behavioral: Flexiquit

INTERVENTIONS:
Behavioral: Flexiquit — Digital avatar-led Acceptance and Commitment Therapy for smoking cessation
  Arms: Flexiquit

SUMMARY:
Smoking remains a global concern, especially for youth where developmentally-suited smoking cessation programs are lacking and especially among those not presenting for treatment on their own. We aimed to assess the effectiveness of an avatar-led digitalized smoking cessation intervention (Flexiquit) based on Acceptance and Commitment Therapy (ACT) for young adult smokers at all levels of motivation to quit.

DETAILED DESCRIPTION:
Cigarette smoking is associated with various health problems, particularly certain forms of cancer and early death (Centers for Disease Control and Prevention, 1997). More recently, smoking has become a global problem among youth and it is imperative that research puts an emphasis on prevention and intervention particularly in this age group (World Health Organization, 2009). Over the past few years, research has shown that internet-based interventions are more cost effective, cater to individuals who are unable/unwilling to attend weekly treatment sessions with a therapist, and are promising in terms of improving attrition rates, a major problem with most treatment trials. Moreover, internet-based interventions use technology often utilized to attract youth (interactive games, animation, video clips etc.) and thus may reach and engage a wider range of individuals than traditional face-to-face interventions. ACT is an empirically-based intervention that uses acceptance and mindfulness strategies and has been shown to increase psychological flexibility. The aim of the present study is to investigate the usefulness and effectiveness of an Acceptance and Commitment Therapy (ACT) internet-based smoking cessation intervention program for college, high school and vocational school student smokers. Findings are expected to show that a digitalized program designed to engage youth in smoking cessation can result in quitting smoking and has a high applicability potential especially among the hard-to-reach population of youth.

ELIGIBILITY:
Inclusion Criteria:

* Regular smoker (at least 1 cigarette per day)
* Parental consent for those under 18years of age

Exclusion Criteria:

* Currently enrolled in another smoking cessation program

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Quit rate | Post-intervention (following completion of digital session 5) and follow-up (3 months and 6 months after post-intervention)
  Change in Smoking quit status at each assessment point
Change in Number of cigarettes | Post-intervention (following completion of digital session 5) and follow-up (3 months and 6 months after post-intervention)
  Change in the number of cigarettes smoked per day

SECONDARY OUTCOMES:
Change in Nicotine Dependence | Post-intervention (following completion of digital session 5) and follow-up (3 months and 6 months after post-intervention)
  Change in the Fagerstrom Test of Nicotine Dependence scores
Change in Readiness to quit | Post-intervention (following completion of digital session 5) and follow-up (3 months and 6 months after post-intervention)
  Change in the Contemplation Ladder assessing stages of change
Change in self-efficacy to not smoke in specific situations | Post-intervention (following completion of digital session 5) and follow-up (3 months and 6 months after post-intervention)
  Change in Smoking Self-Efficacy Questionnaire scores

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cyprus, Nicosia, Non-US/Non-Canadian, Cyprus

IPD SHARING:
Plan to Share IPD: No